CLINICAL TRIAL: NCT06095466
Title: Diagnosis and Pathogenetic Mechanisms in Cirrhotic Cardiomyopathy Based on Point-of-care Echocardiography, Biomarkers and Histology
Brief Title: Cirrhotic Cardiomyopathy Based on Point-of-care Echocardiography, Biomarkers and Histology
Status: Recruiting | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: INT/IEC/2023/SPL-963
Record Dates: First submitted 2023-09-19; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Cirrhotic Cardiomyopathy; Cirrhosis, Liver; Cardiac Disease
MeSH Terms: conditions — Liver Cirrhosis; Heart Diseases | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cirrhotic cardiomyopathy: Cirrhotic cardiomyopathy, among a broad spectrum of cardiac complications in cirrhosis, is characterized by systolic and diastolic cardiac dysfunction and electrocardiographic changes. However, it is seen more in NASH related cirrhotic patients, who have an additional risk of developing cardiac complications. Cirrhosis contributes to a including cirrhotic cardiomyopathy owing to various pathological conditions interlinked at the cellular and molecular level. A hyperdynamic circulatory state caused due to excessive release of vasodilators in a pro-inflammatory condition of cirrhosis, along with negative-inotropic pathways contributes to the development of a compromised cardiac function. Electrocardiography, 2D echocardiography with tissue Doppler or speckle tracking are the routine diagnostic tests used to diagnose CCM.
  Interventions: Device: Echocardiographic assessment; Diagnostic Test: Histopathology and Immunohistochemistry

INTERVENTIONS:
Device: Echocardiographic assessment — M mode, cross sectional and pulsed wave Doppler Echocardiographic examinations will be performed using a with a 2.5 MHz wide angle phased array transducer. Patients will be laid in left lateral position and examined in standard parasternal long and short axis and apical views. Short axis recordings will be performed at the level of the papillary muscles. M mode tracings will be recorded at the level of the papillary muscles and the aortic valves, with 2 -D guidance. LV wall thickness and cavity diameters will be measured by M mode, through the largest diameter of the ventricle, if possible, both in diastole and systole. Using the cross-sectional images as a guide, the M mode tracing of the left ventricle will obtained to calculate measurements according to the recommendations of American Society of Echocardiography.
Diagnostic Test: Histopathology and Immunohistochemistry — In patients who do not survive, we will take a trucut core biopsy from the ventricular myocardium, using ultrasound guidance. Cardiac tissue slices preserve the heterogeneous structure and multicellularity of the myocardium and allow its functional characterization. However, in this protocol, only those patients who consent to autopsy or those who consent to most mortem biopsy will be sampled for cardiac histology in CCM. Thus samples for histology and immunohistopathology will be available in only a few patients.
  For the immunohistochemistry study, the sections will be collected on the poly-L-lysine covered slides and dried in a thermostat, at 37°C, for 24 hours, for increasing the adherence of the biological material to the histological slide.

SUMMARY:
Cirrhotic cardiomyopathy is associated with increased risk of complications like hepatorenal syndrome, refractory ascites, impaired response to stressors including sepsis, bleeding or transplantation, poor health related quality of life and increased morbidity and mortality. Left ventricular diastolic dysfunction (LVDD) is associated with risk of hepatorenal syndrome (HRS) , septic shock. , heart failure in the perioperative period following liver transplantation, and after trans-jugular intrahepatic portosystemic shunt (TIPS) insertion . The echocardiographic E/e' ratio is a predictor of survival in LVDD, with multiple studies, including prospective data from our Centre.

DETAILED DESCRIPTION:
The inability of the heart to cope with stress or sepsis induced circulatory failure is a key concept of the increased mortality risk due to LVDD. In view of the metabolic syndrome and diabetes epidemic and an increasing number of patients being diagnosed with non-alcoholic fatty liver disease, there is increased risk of developing cardiac dysfunction due to multiple comorbidities including coronary artery disease, hypertensive heart disease, cirrhotic cardiomyopathy, which are contributors to overall cardiovascular risk of mortality.

In this project the investigators will screen critically ill patients with cirrhosis admitted to the intensive care unit for presence of cirrhotic cardiomyopathy and perform point-of-care echocardiography, electrocardiography, and cardiorenal biomarker tests for determination of outcomes in CCM. In patients who do not survive, the cardiac histology will be assessed by ultrasound guided myocardial biopsy to assess degree of inflammation and fibrosis in CCM.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis who have been diagnosed by clinical, biochemical, histological (when available) criteria plus ultrasound imaging will be included if they meet the following:

  * Age range of 18-65 years
  * Cirrhosis with critical illness admitted to the Liver Intensive Care Unit

Exclusion Criteria:

* Age >65 years
* Chronic renal disease
* Pregnancy and peripartum cardiomyopathy
* Valvular heart disease
* Sick sinus syndrome/ Pacemaker
* Transjugular intrahepatic porto systemic shunt (TIPS) insertion
* Hepatocellular carcinoma
* Anemia Hb < 8gm/dl in females, and < 9 gm/dl in males at the time of assessment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this study is all critically ill cirrhotic patients admitted to the Liver Intensive Care Unit of the Department of Hepatology, PGIMER Chandigarh
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Determine the prevalence of cirrhotic cardiomyopathy in critically ill patients with cirrhosis | At Enrollment
  CCM is independent of etiology, and all patients should be assessed for this under diagnosed complication of liver disease. The presence of metabolic syndrome, use of alcohol and cirrhosis can contribute synergistically as risk factors for clinically undiagnosed case of CCM. In a nutshell, the cirrhotic heart displays a variation of structure and size, atherosclerotic lesions, and myocardium hypertrophy with impaired functioning, with fibrosis and remodeling in late stages.
  The prevalence of patients with CCM diagnosed as per the 2020 CCM criteria of the AASLD will be assessed.

SECONDARY OUTCOMES:
Determine severity of cardiac dysfunction in critically ill patients with cirrhosis | At Enrollment
  Grade of left ventricular diastolic dysfunction will be assessed. Systolic function including stroke volume, velocity time integral and cardiac index will be assessed.
Determine the POCUS determinants of cardiac dysfunction in critically ill patients with cirrhosis | At Enrollment
  POCUS variables like cardiac output, SVRI, right ventricular variables, pulmonary artery pressure will be recorded.
Determine the cardiac histology changes in critically ill patients with cirrhosis | At the time of demise
  In patients who consent for autopsy or post mortem biopsy, cardiac, liver, renal, lung and splenic histological changes will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Madhumita Premkumar, Sector-12, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Premkumar M, Devurgowda D, Vyas T, Shasthry SM, Khumuckham JS, Goyal R, Thomas SS, Kumar G. Left Ventricular Diastolic Dysfunction is Associated with Renal Dysfunction, Poor Survival and Low Health Related Quality of Life in Cirrhosis. J Clin Exp Hepatol. 2019 May-Jun;9(3):324-333. doi: 10.1016/j.jceh.2018.08.008. Epub 2018 Aug 30. PMID 31360025
- [Background] Premkumar M, Anand AC. Overview of Complications in Cirrhosis. J Clin Exp Hepatol. 2022 Jul-Aug;12(4):1150-1174. doi: 10.1016/j.jceh.2022.04.021. Epub 2022 May 14. PMID 35814522
- [Background] Kaur H, Premkumar M. Diagnosis and Management of Cirrhotic Cardiomyopathy. J Clin Exp Hepatol. 2022 Jan-Feb;12(1):186-199. doi: 10.1016/j.jceh.2021.08.016. Epub 2021 Aug 21. PMID 35068798
- [Background] Izzy M, VanWagner LB, Lin G, Altieri M, Findlay JY, Oh JK, Watt KD, Lee SS; Cirrhotic Cardiomyopathy Consortium. Redefining Cirrhotic Cardiomyopathy for the Modern Era. Hepatology. 2020 Jan;71(1):334-345. doi: 10.1002/hep.30875. Epub 2019 Oct 11. PMID 31342529
- [Background] Wiese S, Voiosu A, Hove JD, Danielsen KV, Voiosu T, Gronbaek H, Moller HJ, Genovese F, Reese-Petersen AL, Mookerjee RP, Clemmesen JO, Gotze JP, Andersen O, Moller S, Bendtsen F. Fibrogenesis and inflammation contribute to the pathogenesis of cirrhotic cardiomyopathy. Aliment Pharmacol Ther. 2020 Jul;52(2):340-350. doi: 10.1111/apt.15812. Epub 2020 Jun 11. PMID 32524673